CLINICAL TRIAL: NCT04562597
Title: A Pilot Trial to Determine the Effective Dose of N-acetylcysteine for Opioid Reduction in Patients Undergoing Spine Surgery.
Brief Title: A Pilot Trial to Determine the Effective N-acetylcysteine Dose for Opioid Reduction for Spine Surgery.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Sylvia Wilson, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00099062
Record Dates: First submitted 2020-09-10; First posted 2020-09-24 (Actual); Results first posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Surgery

STUDY DESIGN:
Intervention Model Description: PHASE I. First 20 subjects (4 arms): We will initially randomize 5 patients to each dose group (placebo, 50, 100, and 150 mg/kg) to estimate the dose response curve and to identify the optimal dose. After enrollment of the first 20 patients, the study will undergo review by the study team and statistician.
  PHASE II: (2 arms) If the dose response curve is adequate and the optimal dose identified, 15 additional participants will be randomized to placebo and 15 to the optimal dose to estimate the difference in opioid consumption between patients on placebo vs. the optimal dose.
  Primary and secondary outcomes will be evaluated only for the placebo and optimal NAC groups.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Dose Response Curve Placebo (Placebo Comparator): 5 participants will be randomized to the placebo group to estimate the dose response curve and to identify the optimal dose.
  Interventions: Drug: Dose Response Curve Placebo
- Dose Response Curve N-acetylcysteine 50 mg/kg (Active Comparator): 5 participants will be randomized to the N-acetylcysteine 50 mg/kg group to estimate the dose response curve and to identify the optimal dose.
  Interventions: Drug: Dose Response Curve N-acetylcysteine 50 mg/kg
- Dose Response Curve N-acetylcysteine 100 mg/kg (Active Comparator): 5 participants will be randomized to the N-acetylcysteine 100 mg/kg group to estimate the dose response curve and to identify the optimal dose.
  Interventions: Drug: Dose Response Curve N-acetylcysteine 100 mg/kg
- Dose Response Curve N-acetylcysteine 150 mg/kg (Active Comparator): 5 participants will be randomized to the N-acetylcysteine 150 mg/kg group to estimate the dose response curve and to identify the optimal dose.
  Interventions: Drug: Dose Response Curve N-acetylcysteine 150 mg/kg
- Opioid Reduction with Optimal N-acetylcysteine Dose (Active Comparator): Once the optimal N-acetylcysteine dose is identified, 15 additional participants will be randomized to the optimal dose to estimate the difference in opioid consumption between patients on placebo vs. the optimal dose. Primary and secondary outcomes will only be evaluated for the placebo group and optimal NAC group.
  Interventions: Drug: Opioid Reduction with Optimal N-acetylcysteine Dose
- Placebo (Placebo Comparator): 15 Participants will be randomized to placebo to estimate the difference in opioid consumption between patients on placebo vs. the optimal dose. Primary and secondary outcomes will only be evaluated for the placebo group and optimal NAC group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dose Response Curve Placebo — 5 participants will be randomized to the placebo group to estimate the dose response curve and to identify the optimal dose.
  Arms: Dose Response Curve Placebo
Drug: Dose Response Curve N-acetylcysteine 50 mg/kg — 5 participants will be randomized to the N-acetylcysteine 50 mg/kg group to estimate the dose response curve and to identify the optimal dose.
  Arms: Dose Response Curve N-acetylcysteine 50 mg/kg
Drug: Dose Response Curve N-acetylcysteine 100 mg/kg — 5 participants will be randomized to the N-acetylcysteine 100 mg/kg group to estimate the dose response curve and to identify the optimal dose.
  Arms: Dose Response Curve N-acetylcysteine 100 mg/kg
Drug: Dose Response Curve N-acetylcysteine 150 mg/kg — 5 participants will be randomized to the N-acetylcysteine 150 mg/kg group to estimate the dose response curve and to identify the optimal dose.
  Arms: Dose Response Curve N-acetylcysteine 150 mg/kg
Drug: Opioid Reduction with Optimal N-acetylcysteine Dose — Once the optimal N-acetylcysteinedose is identified, 15 participants will be randomized to the optimal dose (50,100, or 150 mg/kg) to estimate the difference in opioid consumption between patients administered optimal N-acetylcysteine dose or placebo.
  Arms: Opioid Reduction with Optimal N-acetylcysteine Dose
Drug: Placebo — 15 Participants will be randomized to placebo to estimate the difference in opioid consumption between patients administered optimal N-acetylcysteine dose or placebo.
  Arms: Placebo

SUMMARY:
Determine the optimal dose of IV N-acetylcysteine (NAC) to produce opioid reduction following spine surgery and estimate the difference in opioid consumption between placebo and the selected optimal dose.

DETAILED DESCRIPTION:
First 20 subjects: 5 participants will be randomized to each dose group (placebo, 50, 100, and 150 mg/kg) to estimate the dose response curve and to identify the optimal dose.

If the dose response curve is adequate and the optimal dose identified, 15 additional participants will be randomized to placebo and 15 to the optimal dose to estimate the difference in opioid consumption between participants on placebo vs. the optimal dose. (Total of 50 subjects with 20 from dose response curve and 30 to estimate the difference in opioid consumption.)

If the dose response curve is not adequate after the initial 20 subjects 5 per each dose group, then an additional 5 participants will be randomized and to each dose group (placebo, 50, 100, and 150 mg/kg) to estimate the dose response curve and to identify the optimal dose. Once the optimal dose is identified with these initial 40 patients, 10 additional participants will be randomized to placebo and 10 to the optimal dose to estimate the difference in opioid consumption between participants on placebo vs. the optimal dose. (60 patients total with 40 to create the dose response curve and 20 more to estimate the difference in opioid consumption.)

A sample size of 20 subjects per group (placebo and optimal dose) allows us to estimate a 95% confidence interval for the mean difference in opioid consumption with a width of + 0.64 standard deviations from the mean. 70 subjects may be enrolled to account for withdrawal but the study will be completed once 50 or 60 subjects (based on the number of subjects required to create the dose response curve) have completed the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective spine surgery involving 4 levels or less of the thoracic, lumbar, or sacral spine.
* 18 years of age and older.

Exclusion Criteria:

* Less than 40kg in weight.
* Unable to provide written, informed consent.
* History of an adverse or anaphylactoid reaction to acetylcysteine.
* Active asthma, wheezing, or using inhaled bronchodilators.
* Pregnant Women
* Known blood clotting deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Wilson, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hall AJ, Logan JE, Toblin RL, Kaplan JA, Kraner JC, Bixler D, Crosby AE, Paulozzi LJ. Patterns of abuse among unintentional pharmaceutical overdose fatalities. JAMA. 2008 Dec 10;300(22):2613-20. doi: 10.1001/jama.2008.802. PMID 19066381
- [Background] Pieralisi A, Martini C, Soto D, Vila MC, Calvo JC, Guerra LN. N-acetylcysteine inhibits lipid accumulation in mouse embryonic adipocytes. Redox Biol. 2016 Oct;9:39-44. doi: 10.1016/j.redox.2016.05.006. Epub 2016 May 27. PMID 27281491
- [Background] Heim MU, Alraun K, Leeping M, Schwarzfischer G, Bock M, Kling A, Mempel W. [Incidence of the detection of erythrocyte antibodies in relation to screening test cells]. Beitr Infusionsther. 1992;30:443-5. German. PMID 1284756
- [Background] Guo F, Li Y, Wang J, Li Y, Li Y, Li G. Stanniocalcin1 (STC1) Inhibits Cell Proliferation and Invasion of Cervical Cancer Cells. PLoS One. 2013;8(1):e53989. doi: 10.1371/journal.pone.0053989. Epub 2013 Jan 29. PMID 23382863
- [Background] Bavarsad Shahripour R, Harrigan MR, Alexandrov AV. N-acetylcysteine (NAC) in neurological disorders: mechanisms of action and therapeutic opportunities. Brain Behav. 2014 Mar;4(2):108-22. doi: 10.1002/brb3.208. Epub 2014 Jan 13. PMID 24683506
- [Background] Tardiolo G, Bramanti P, Mazzon E. Overview on the Effects of N-Acetylcysteine in Neurodegenerative Diseases. Molecules. 2018 Dec 13;23(12):3305. doi: 10.3390/molecules23123305. PMID 30551603
- [Background] Monti DA, Zabrecky G, Kremens D, Liang TW, Wintering NA, Bazzan AJ, Zhong L, Bowens BK, Chervoneva I, Intenzo C, Newberg AB. N-Acetyl Cysteine Is Associated With Dopaminergic Improvement in Parkinson's Disease. Clin Pharmacol Ther. 2019 Oct;106(4):884-890. doi: 10.1002/cpt.1548. Epub 2019 Jul 17. PMID 31206613
- [Background] Monti DA, Zabrecky G, Kremens D, Liang TW, Wintering NA, Cai J, Wei X, Bazzan AJ, Zhong L, Bowen B, Intenzo CM, Iacovitti L, Newberg AB. N-Acetyl Cysteine May Support Dopamine Neurons in Parkinson's Disease: Preliminary Clinical and Cell Line Data. PLoS One. 2016 Jun 16;11(6):e0157602. doi: 10.1371/journal.pone.0157602. eCollection 2016. PMID 27309537
- [Background] Holmay MJ, Terpstra M, Coles LD, Mishra U, Ahlskog M, Oz G, Cloyd JC, Tuite PJ. N-Acetylcysteine boosts brain and blood glutathione in Gaucher and Parkinson diseases. Clin Neuropharmacol. 2013 Jul-Aug;36(4):103-6. doi: 10.1097/WNF.0b013e31829ae713. PMID 23860343
- [Background] Coles LD, Tuite PJ, Oz G, Mishra UR, Kartha RV, Sullivan KM, Cloyd JC, Terpstra M. Repeated-Dose Oral N-Acetylcysteine in Parkinson's Disease: Pharmacokinetics and Effect on Brain Glutathione and Oxidative Stress. J Clin Pharmacol. 2018 Feb;58(2):158-167. doi: 10.1002/jcph.1008. Epub 2017 Sep 22. PMID 28940353
- [Background] Halboub E, Alkadasi B, Alakhali M, AlKhairat A, Mdabesh H, Alkahsah S, Abdulrab S. N-acetylcysteine versus chlorhexidine in treatment of aphthous ulcers: a preliminary clinical trial. J Dermatolog Treat. 2021 Sep;32(6):649-653. doi: 10.1080/09546634.2019.1688231. Epub 2019 Nov 21. PMID 31679408
- [Background] Li J, Xu L, Deng X, Jiang C, Pan C, Chen L, Han Y, Dai W, Hu L, Zhang G, Cheng Z, Liu W. N-acetyl-cysteine attenuates neuropathic pain by suppressing matrix metalloproteinases. Pain. 2016 Aug;157(8):1711-1723. doi: 10.1097/j.pain.0000000000000575. PMID 27075430
- [Background] Notartomaso S, Scarselli P, Mascio G, Liberatore F, Mazzon E, Mammana S, Gugliandolo A, Cruccu G, Bruno V, Nicoletti F, Battaglia G. N-Acetylcysteine causes analgesia in a mouse model of painful diabetic neuropathy. Mol Pain. 2020 Jan-Dec;16:1744806920904292. doi: 10.1177/1744806920904292. PMID 32009537
- [Background] Dludla PV, Nkambule BB, Dias SC, Johnson R. Cardioprotective potential of N-acetyl cysteine against hyperglycaemia-induced oxidative damage: a protocol for a systematic review. Syst Rev. 2017 May 12;6(1):96. doi: 10.1186/s13643-017-0493-8. PMID 28499416
- [Background] Hoffer BJ, Pick CG, Hoffer ME, Becker RE, Chiang YH, Greig NH. Repositioning drugs for traumatic brain injury - N-acetyl cysteine and Phenserine. J Biomed Sci. 2017 Sep 9;24(1):71. doi: 10.1186/s12929-017-0377-1. PMID 28886718
- [Background] Howard RJ, Blake DR, Pall H, Williams A, Green ID. Allopurinol/N-acetylcysteine for carbon monoxide poisoning. Lancet. 1987 Sep 12;2(8559):628-9. doi: 10.1016/s0140-6736(87)93018-2. No abstract available. PMID 2887913
- [Background] Hamamsy ME, Bondok R, Shaheen S, Eladly GH. Safety and efficacy of adding intravenous N-acetylcysteine to parenteral L-alanyl-L-glutamine in hospitalized patients undergoing surgery of the colon: a randomized controlled trial. Ann Saudi Med. 2019 Jul-Aug;39(4):251-257. doi: 10.5144/0256-4947.2019.251. Epub 2019 Aug 5. PMID 31381364
- [Background] Soleimani A, Habibi MR, Hasanzadeh Kiabi F, Alipour A, Habibi V, Azizi S, Emami Zeydi A, Sohrabi FB. The effect of intravenous N-acetylcysteine on prevention of atrial fibrillation after coronary artery bypass graft surgery: a double-blind, randomised, placebo-controlled trial. Kardiol Pol. 2018;76(1):99-106. doi: 10.5603/KP.a2017.0183. Epub 2017 Oct 5. PMID 28980294
- [Background] Sins JWR, Fijnvandraat K, Rijneveld AW, Boom MB, Kerkhoffs JH, van Meurs AH, de Groot MR, Heijboer H, Dresse MF, Le PQ, Hermans P, Vanderfaeillie A, Van Den Neste EW, Benghiat FS, Kesse-Adu R, Delannoy A, Efira A, Azerad MA, de Borgie CA, Biemond BJ. Effect of N-acetylcysteine on pain in daily life in patients with sickle cell disease: a randomised clinical trial. Br J Haematol. 2018 Aug;182(3):444-448. doi: 10.1111/bjh.14809. Epub 2017 Jun 23. No abstract available. PMID 28643376
- [Background] Heidari N, Sajedi F, Mohammadi Y, Mirjalili M, Mehrpooya M. Ameliorative Effects Of N-Acetylcysteine As Adjunct Therapy On Symptoms Of Painful Diabetic Neuropathy. J Pain Res. 2019 Nov 19;12:3147-3159. doi: 10.2147/JPR.S228255. eCollection 2019. PMID 31819599
- [Background] Kerr F, Dawson A, Whyte IM, Buckley N, Murray L, Graudins A, Chan B, Trudinger B. The Australasian Clinical Toxicology Investigators Collaboration randomized trial of different loading infusion rates of N-acetylcysteine. Ann Emerg Med. 2005 Apr;45(4):402-8. doi: 10.1016/j.annemergmed.2004.08.040. PMID 15795719
- [Background] Yip L, Dart RC. A 20-hour treatment for acute acetaminophen overdose. N Engl J Med. 2003 Jun 12;348(24):2471-2. doi: 10.1056/NEJM200306123482422. No abstract available. PMID 12802041
- [Derived] Wilson SH, Sirianni JM, Bridges KH, Wolf BJ, Valente IE, Scofield MD. The impact of intraoperative N-acetylcysteine on opioid consumption following spine surgery: a randomized pilot trial. Pain Manag. 2023 Oct;13(10):593-602. doi: 10.2217/pmt-2023-0061. Epub 2023 Oct 25. PMID 37877260

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1: NAC (0mg/kg): (n=5) 5 participants randomized to the placebo group to estimate the dose response curve and to identify the optimal dose.
- Period 1: NAC (50mg/kg): (n=5) 5 participants will be randomized to the N-acetylcysteine 50 mg/kg group to estimate the dose response curve and to identify the optimal dose.
- Period 1: NAC (100mg/kg): (n=5) 5 participants will be randomized to the N-acetylcysteine 100 mg/kg group to estimate the dose response curve and to identify the optimal dose.
- Period 1: NAC (150mg/kg): (n=5) 5 participants will be randomized to the N-acetylcysteine 150 mg/kg group to estimate the dose response curve and to identify the optimal dose.
- Period 2: NAC (0mg/kg): (n=15) 15 additional participants randomized to placebo
- Period 2: NAC (150mg/kg): (n=15) Since optimal not identified with dose response curve, 15 more subjects enrolled in 150 mg/kg group for final comparison with placebo.
Period: Overall Study
Arm/Group | Period 1: NAC (0mg/kg) | Period 1: NAC (50mg/kg) | Period 1: NAC (100mg/kg) | Period 1: NAC (150mg/kg) | Period 2: NAC (0mg/kg) | Period 2: NAC (150mg/kg)
Started | 5 | 5 | 5 | 5 | 15 | 15
Completed | 5 | 5 | 5 | 5 | 15 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- NAC (0mg/kg): (n=20) 5 participants randomized to the placebo group to estimate the dose response curve and to identify the optimal dose. Then 15 more patients enrolled for final comparison versus optimal dose.
- NAC (50mg/kg): (n=5) 5 participants will be randomized to the N-acetylcysteine 50 mg/kg group to estimate the dose response curve and to identify the optimal dose.
- NAC (100mg/kg): (n=5) 5 participants will be randomized to the N-acetylcysteine 100 mg/kg group to estimate the dose response curve and to identify the optimal dose.
- NAC (150mg/kg): (n=20) 5 participants will be randomized to the N-acetylcysteine 150 mg/kg group to estimate the dose response curve and to identify the optimal dose. Since optimal not identified with dose response curve, 15 more subjects enrolled in 150 mg/kg group for final comparison with placebo.
- Total: Total of all reporting groups
Arm/Group | NAC (0mg/kg) | NAC (50mg/kg) | NAC (100mg/kg) | NAC (150mg/kg) | Total
Number analyzed (Participants) | 20 | 5 | 5 | 20 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (12.8) | 68.4 (8.21) | 71.6 (7.54) | 67.4 (6.62) | 64.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 2 | 7 | 20
  Male | 11 | 3 | 3 | 13 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 0 | 4 | 10
  White | 15 | 3 | 5 | 16 | 39
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 5 | 5 | 20 | 50
Home opioid use (yes) [Number; unit: participants] | 5 | 2 | 1 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption 12 Hours Post Operative
Description: Post operative opioid consumption in the 12 hours that occur post-operatively.
Time Frame: 12 hours
Population: Primary and secondary outcomes were only be evaluated for the placebo and optimal NAC groups. Data are reported as mean (95% CI) estimated from a linear mixed model of opioid consumption over time including main effects for treatment group, postoperative time, and the interaction between treatment group and postoperative time and a random subject effect.
Measure: Mean (95% Confidence Interval); unit: IV morphine mg equivalents
Groups:
- Placebo: NAC 0 mg/kg
- N-acetylcysteine (NAC): N-acetylcysteine (NAC)150 mg/kg
Arm/Group | Placebo | N-acetylcysteine (NAC)
Number analyzed (Participants) | 20 | 20
IV morphine mg equivalents | 19.4 [10.8 to 28] | 15.6 [7.02 to 24.2]

2. Secondary Outcome: Opioid Consumption Every 6 Hours Post Operative
Description: Post operative opioid consumption ry 6 hours post operative. Data are reported as mean (95% CI) or mean difference (95% CI) estimated from a linear mixed model of opioid consumption over time including main effects for treatment group, postoperative time, and the interaction between treatment group and postoperative time and a random subject effect.
Time Frame: 6-48 hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: IV morphine mg equivalents
Groups:
- N-acetylcysteine (NAC): N-acetylcysteine (NAC) 150 mg/kg
Arm/Group | Placebo | N-acetylcysteine (NAC)
Number analyzed (Participants) | 20 | 20
IV morphine mg equivalents
  6 hours | 14.6 [5.97 to 23.1] | 12.0 [3.43 to 20.6]
  18 hours | 25.0 [16.4 to 33.6] | 19.9 [11.3 to 28.5]
  24 hours | 29.6 [21.0 to 38.2] | 24.7 [16.2 to 33.3]
  30 hours | 34.0 [25.4 to 42.6] | 27.2 [18.7 to 35.8]
  36 hours | 37.9 [29.4 to 46.5] | 29.7 [21.1 to 38.3]
  42 | 40.9 [32.3 to 49.5] | 33.1 [24.5 to 41.7]
  48 | 43.3 [34.7 to 51.0] | 34.9 [26.4 to 43.6]

ADVERSE EVENTS:
Time Frame: 48 hours
Groups:
- Placebo: N-acetylcysteine (NAC) 0 mg/kg
- NAC 50 mg/kg: N-acetylcysteine (NAC) 50 mg/kg
- NAC 100 mg/kg: N-acetylcysteine (NAC) 100 mg/kg
- NAC 150 mg/kg: N-acetylcysteine (NAC) 150 mg/kg
Arm/Group | Placebo | NAC 50 mg/kg | NAC 100 mg/kg | NAC 150 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/5 | 0/5 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/5 | 0/5 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/5 | 0/5 | 0/20

LIMITATIONS AND CAVEATS:
* Opioid consumption was highly variable. This is likely due to the small sample size.
* Data only collected up to 48 hours postoperative, and this limits our ability to comment more on the usefulness of NAC as an agent for patients with chronic pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT04562597/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT04562597/SAP_001.pdf